CLINICAL TRIAL: NCT06839079
Title: Feasibility RCT of an Adapted Cognitive Rehabilitation Program for Refugees and Asylum Seekers With TBI and Cognitive Impairment
Brief Title: Cognitive Rehabilitation for Refugees With Traumatic Brain Injury and Cognitive Impairment
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Collaborators: National Institute of Neurological Disorders and Stroke (NINDS) (NIH)
Responsible Party: Principal Investigator, Altaf Saadi, MD MSc, Associate Professor of Neurology, Massachusetts General Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Health Services Research
Other Study IDs: 2024P002728; K23NS128164 (NIH)
Record Dates: First submitted 2025-02-04; First posted 2025-02-21 (Actual); Last update posted 2025-10-29 (Actual); Status verified 2025-10

CONDITIONS: TBI (Traumatic Brain Injury); Cognitive Symptoms
Keywords: Traumatic Brain Injury; Cognition; Refugees; Asylum Seekers
MeSH Terms: conditions — Brain Injuries, Traumatic; Neurobehavioral Manifestations

STUDY DESIGN:
Intervention Model Description: Participants will be randomly assigned to one of two groups:
  Group A will receive the intervention immediately. Group B will initially not receive the intervention (waitlist control). After approximately 12 weeks period, Group B will receive the intervention (delayed start).
  All participants will complete questionnaires at three time points:
  Baseline (after enrollment) Approximately 12 weeks after baseline. Approximately 24 weeks after baseline.
Who Masked: Investigator, Outcomes Assessor
Masking Description: The investigator and members of the study staff conducting assessments will be blinded to participant's group assignment.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Adapted cognitive rehabilitation program intervention (Experimental): Those in the immediate intervention arm will receive the adapted cognitive rehabilitation therapy program which includes virtual sessions delivered by a paraprofessional focused on improving cognitive function. They will complete baseline assessments (target outcomes and demographic and general health information) and take part in the post-intervention assessments (target outcomes and feasibility, acceptability, and satisfaction measures) at approximately 12 weeks and 24 weeks after baseline.
  Interventions: Behavioral: A Trauma-informed, Paraprofessional Delivered Virtual Cognitive Rehabilitation Program
- Waitlist Control (No Intervention): Those in the waitlist control arm will complete baseline assessments (target outcomes and demographic and health information) and receive communications once a week mimicking the contact of the intervention. They will also participate in the post-assessment at approximately 12 weeks, after which they will receive the intervention. After that, they will complete the third assessment, at approximately 24 weeks (target outcomes and feasibility, acceptability, and satisfaction measures)

INTERVENTIONS:
Behavioral: A Trauma-informed, Paraprofessional Delivered Virtual Cognitive Rehabilitation Program — The intervention will involve 8 proposed individual sessions conducted virtually by a trained bilingual paraprofessional. The intervention will be provided in English or Spanish depending on the participant's preference. The sessions cover psychoeducation about TBI and related symptoms like depression and anxiety, and cognitive activities to address cognitive symptoms (e.g., relaxation strategies and exercises around improving attention, concentration, learning, and memory). Each session covers the topic, real-life examples and practice, and exercises to do outside of the sessions.
  Arms: Adapted cognitive rehabilitation program intervention

SUMMARY:
Researchers at Massachusetts General Hospital are looking to see if a program created to help improve thinking and memory can work for refugees with traumatic brain injury (TBI). They're checking if this program is practical and if people find it helpful.

The study will have two groups. Participants will complete a first questionnaire and then be assigned to a group by chance. One group will participate in the program immediately and then answer the second questionnaire (approximately 3 months after the first questionnaire they did). Then they will wait and then answer the third and final questionnaire approximately 6 months after the first one.

The second group will wait and answer the second questionnaire approximately 3 months after the first one. Then they will receive the program and answer the third and final questionnaire (approximately 6 months after the first one they did.)

DETAILED DESCRIPTION:
There are many refugees and asylum seekers in the world ("refugees" from here on for simplicity). Many of them have suffered from traumatic brain injury (TBI) as a result of traumatic experiences like torture and interpersonal violence. Because of one or more TBI's, they can experience cognitive issues, or issues with learning, thinking, concentration and memory. Cognitive rehabilitation can be one effective way to reduce the burden of cognitive issues following TBI. Cognitive rehabilitation refers to a functionally oriented service of cognitive activities that can aim to lessen cognitive impairments or lessen the disabling impact of these impairments. Yet not all people access cognitive rehabilitation equally. We have tailored an existing cognitive rehabilitation program to be delivered virtually and through a paraprofessional for refugees with TBI and cognitive issues. A paraprofessional refers to a person from the community who does not have specialized medical training.

This is a pilot feasibility randomized trial where English and Spanish-speaking participants will be randomized to either the adapted intervention (n = 25) or a wait-list control (n = 25) in the first stage. The participants in the adapted intervention will receive the intervention first while people in the wait-list control wait. People in the waitlist control will receive the intervention after approximately 12 weeks. All participants will have assessments at baseline, approximately 12 weeks, and 24 weeks after baseline.

During the intervention, participants will complete a program that involves 8 sessions. The sessions will cover material relating to cognitive rehabilitation, such as exercises relating to external or internal memory strategies, aimed to improve cognitive challenges people with TBI experience.

Participants assigned to the immediate intervention will receive the program and then answer the second questionnaire, approximately 12-weeks after their baseline. They will complete the third questionnaire approximately 24-weeks after their baseline

Participants assigned to the waitlist control group will answer the baseline and second questionnaire 12 weeks after. They will then receive the intervention and complete the third questionnaire, approximately 24-weeks after their baseline.

ELIGIBILITY:
Inclusion Criteria:

1. Identify as an asylum seeker, refugee or have been granted asylum or other form of humanitarian relief.
2. Mild or moderate TBI sustained after the age of 18
3. Age 18-65
4. Subjective cognitive impairment
5. English or Spanish language proficiency
6. Ability to provide verbal informed consent
7. Ability and willingness to answer questionnaires and participation in the Intervention

Exclusion Criteria:

1. Participation in cognitive rehabilitation treatment current or in past 3 months
2. Severe TBI or TBI only sustained under the age of 18
3. Diagnosis of bipolar, psychosis, active substance use, self-reported current active suicidal ideation or plan

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2025-10-15 (Actual); Primary Completion 2027-03 (Estimated); Study Completion 2027-12 (Estimated)

PRIMARY OUTCOMES:
Acceptability of the intervention | Through Intervention participation, an average of 8 weeks, and at the 12 weeks and 24 weeks follow-up questionnaires.
  At least 70% of participants will complete 7 or more sessions. At least 70% of participants will complete their homework. At least 80% of participants will complete the study and 12 weeks assessment. At least 60% of participants will complete the 24 weeks assessment.
Acceptability of the intervention | After the intervention at the 12 weeks and 24 weeks follow-up questionnaires.
  At least 70% of participants will score over the midpoint in the 4-item Acceptability of Intervention Measure. The AIM scale values range from 1 to 5 with a higher score of 20. Higher scores indicate greater acceptability.
Feasibility of the intervention | Baseline, and through Intervention participation, an average of 8 weeks.
  At least 80% of people approached will agree to participate (feasibility of recruitment).
  At least 70% of participants will have no measures fully missing (feasibility of assessments).
Feasibility of the intervention | After the intervention at 12 weeks and 24 weeks follow-up questionnaires.
  At least 70% of participants will score over the midpoint in the 4-item Feasibility of Intervention Measure (FIM). The FIM is a scale whose values range from 1-5 and a higher score of 20. Higher scores indicate greater acceptability.
Satisfaction with the intervention | After the intervention at the, 12 weeks and 24 weeks follow-up questionnaires.
  At least 70% of participants will score over the midpoint in the Client Satisfaction Questionnaire (CSQ-8). Scores for the CSQ-8 range from 8 to 32 and higher scores indicate greater satisfaction.

SECONDARY OUTCOMES:
Potential effectiveness on reducing cognitive impairment symptoms in objective measures | Baseline, 12 weeks and 24 weeks follow-up questionnaires
  Improvement in cognitive function will be assessed through changes on Montreal Cognitive Assessment (MoCA). The MoCA's highest possible score is 30; a score of 26 and higher is considered normal and lower than this cut off will indicate possible cognitive impairment
Potential effectiveness on reducing cognitive impairment symptoms in objective measures | Baseline, 12 weeks and 24 weeks follow-up questionnaires
  Improvement in cognitive function will be assessed through changes on:
  Rowland Universal Dementia Assessment Scale (RUDAS) measure. The RUDAS maximum score is 30; a score of 23 and higher is considered normal and lower than this cut off will indicate possible cognitive impairment.
Potential effectiveness on reducing cognitive impairment symptoms in subjective measures | Baseline, 12 weeks and 24 weeks follow-up questionnaires
  Improvement in cognitive function will be assessed through changes in:
  PROMIS (Patient Reported Outcome Measurement Information System) Short Form v2.0 - Cognitive Function 8a scale. The scale uses a T score metric where 50 is the mean (the average for the United States general population) and 10 is the standard deviation above or below the mean. A higher score indicates better cognitive performance.
Potential effectiveness on reducing cognitive impairment symptoms in subjective measures | Baseline, 12 weeks and 24 weeks follow-up questionnaires
  Improvement in cognitive function will be assessed through changes in the cognitive questions of Neurobehavioral Symptom Inventory (NSI). The NSI total score ranges from 0 to 88 and it can provide raw scores for four domains, one of them cognitive. A higher score indicates more severe post-concussive symptoms.
Potential effectiveness on reducing post-concussive symptoms | Baseline, 12 weeks and 24 weeks follow-up questionnaires
  Improvement in post-concussive symptoms will be measured using the Neurobehavioral Symptom Inventory (NSI). The NSI total score ranges from 0 to 88. A higher score indicates more severe post-concussive symptoms.

CONTACTS AND LOCATIONS:
Locations (1):
- Massachusetts General Hospital, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: Yes
All of individual participant data collected during the trial, after deidentification
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: All data will be made available immediately following first publication relating to clinical trial. No end date.
Access Criteria: Anyone who wishes to access the data will be able to do so from Harvard Dataverse. Data will be stored in accessible formats, such as excel/csv format.

REFERENCES:
- [Background] Parvez A, Percac-Lima S, Saadi A. The Presence and Profile of Neurological Conditions and Associated Psychiatric Comorbidities in U.S. Resettled Refugees: A Retrospective Single Center Study. J Immigr Minor Health. 2023 Apr;25(2):365-373. doi: 10.1007/s10903-022-01409-6. Epub 2022 Oct 17. PMID 36251204
- [Background] Sherman Rosa S, Nadal R, Saadi A. Research Letter: Assessing Traumatic Brain Injury in Refugees: Feasibility, Usability, and Prevalence Insights From a US-Based Clinical Sample. J Head Trauma Rehabil. 2025 Jul-Aug 01;40(4):E334-E339. doi: 10.1097/HTR.0000000000001037. Epub 2025 Jul 1. PMID 39874279
- [Background] Saadi A, Williams J, Parvez A, Alegria M, Vranceanu AM. Head Trauma in Refugees and Asylum Seekers: A Systematic Review. Neurology. 2023 May 23;100(21):e2155-e2169. doi: 10.1212/WNL.0000000000207261. Epub 2023 Apr 5. PMID 37019660
- [Background] Saadi A, Asfour J, Vassimon De Assis M, Wilson T, Haar RJ, Heisler M. Head Injury and Associated Sequelae in Individuals Seeking Asylum in the United States: A Retrospective Mixed-Methods Review of Medico-Legal Affidavits. Brain Sci. 2024 Jun 14;14(6):599. doi: 10.3390/brainsci14060599. PMID 38928599
- [Background] Jahan N, Velasco M, Vranceanu AM, Alegria M, Saadi A. Clinician perspectives on characteristics and care of traumatic brain injury among asylum seekers and refugees. Disabil Rehabil. 2025 Feb;47(3):666-675. doi: 10.1080/09638288.2024.2356014. Epub 2024 Jun 3. PMID 38831593